CLINICAL TRIAL: NCT06708780
Title: Clinical Safety and Therapeutic Effects of Autologous Tregs in T1DM
Brief Title: Immunotherapy with Autologous Tregs in T1DM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Zhu DaLong, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-427-TREG
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treg Group (Experimental): Participants in this group are transplanted with expanded autologous Tregs in addition to routine therapy for T1DM.
  Interventions: Biological: Ex vivo Expanded Human Autologous Regulatory T Cells; Other: Routine Care
- Control Group (Other): Participants in this group receive only routine therapy for T1DM.
  Interventions: Other: Routine Care

INTERVENTIONS:
Biological: Ex vivo Expanded Human Autologous Regulatory T Cells — Peripheral blood component donation is used to collect Treg cells for ex vivo expansion, with technical guidance provided by the Center for Biotechnology Drug Development at the Shanghai Institute of Materia Medica, Chinese Academy of Sciences.
  Arms: Treg Group
Other: Routine Care — Routine care is provided to all participants according to clinical guidelines for T1DM.

SUMMARY:
Type 1 diabetes (T1D) is an autoimmune disease characterized by a progressive immune distruction of pancreat beta cells and deterioration of endogenous insulin secretion. Regulatory T cells (Treg) are fuctionally deficient in T1D, leading to the loss of immune tolerance to the islets and the initiation of an autoimmune attack. Previouse studies have revealed the potential theraputic effects of autologous Treg transplantation in T1D. We have modified the preparation protocol for autologous Tregs. The purpose of this study is to assess the safety and effect of autologous Treg therapy in patients with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of T1DM based on the 2021 version of the Chinese Guidelines for Diagnosis and Treatment of Type 1 Diabetes;
* Aged 8 to 65 years;
* At least one islet autoantibody positive and/or fasting C-peptide does not exceed 300pmol/L;
* Must be capable of providing written, signed, and dated informed consent and willing to comply with research requirements in the study.

Exclusion Criteria:

* The condition of diabetic ketoacidosis has not been controlled;
* Severe allergic constitution;
* Known or suspected tumor;
* Acute pancreatitis, and severe heart, liver, kidney, rheumatic immune, respiratory, nervous or infectious diseases.
* Suffering from gestational diabetes mellitus, single gene mutation diabetes mellitus, diabetes mellitus caused by pancreatic damage or other secondary diabetes mellitus (such as diabetes mellitus caused by Cushing's syndrome, thyroid dysfunction or acromegaly, etc.);
* Women who are pregnant or have a pregnancy plan before and after treatment, and women who are breastfeeding.
* Mental illness, alcohol or drug abuse, unable to cooperate with treatment;
* According to the judgment of the investigator, there are other clinical conditions that may endanger the safety of the subjects.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse events, laboratory abnormalities and other signs of toxicity. | From enrollment to the end of treatment at 1 year

SECONDARY OUTCOMES:
Therapeutic effects on diabetes-related outcomes | From enrollment to the end of treatment at 1 year
  Therapeutic effects on diabetes-related outcomes 1 year after intervention include: 1) C-peptide response during mixed meal tolerance test, reported as the change from baseline in the fasting level, postprandial level and area under the curve; 2) Insulin Use; 3) Hemoglobin A1c.

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Endocrinology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No